CLINICAL TRIAL: NCT04105764
Title: Deep Neuromuscular Blockade to Improve Postoperative Quality of Recovery in Ambulatory Gynaecologic Laparoscopy
Brief Title: Deep NMB in Ambulatory Gynecological Laparoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wahba bakhet (Other)
Collaborators: Elite medical center (Unknown)
Responsible Party: Sponsor-Investigator, Wahba bakhet, LECTRURE, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: elite NMB
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Rocuronium; Neuromuscular Blocking Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEEP BLOCK (Active Comparator): In the deep NMB-group, a PTC of 1 to 2 twitches was maintained, and NMB was reversed with sugammadex at the end of surgery.
  Interventions: Drug: Rocuronium
- Moderate block (Active Comparator): In the moderate NMB group, a TOF count of 1 to 2 was maintained and NMB was reversed with a combination of neostigmine and glycopyrolate at the end of surgery.
  Interventions: Drug: Rocuronium bromide

INTERVENTIONS:
Drug: Rocuronium — DEEP block to PTC 1-3
  Other Names: Neuromuscular blocker
  Arms: DEEP BLOCK
Drug: Rocuronium bromide — MODERATE block to TOF1-2
  Other Names: Neuromuscular blocker
  Arms: Moderate block

SUMMARY:
Gynecological laparoscopic surgery is commonly performed as an ambulatory basis for the aim of rapid discharge, reduce hospital stay with reduced costs and to improve postoperative QOR [1,2]. However, the creation of pneumoperitoneum during laparoscopy may cause postoperative pain and other physiological changes [3], which could influence the postoperative QOR negatively [4]. Poor postoperative QOR leads to prolonged hospital stay [5].

DETAILED DESCRIPTION:
Deep NMB is known to improve surgical conditions and pneumoperitoneium related complications in laparoscopic surgery [6,7,8,9]. However, it is unknown whether deep NMB improves postoperative QOR in ambulatory gynecological laparoscopy.

Therefore, we designed a double blind randomised trial to compare the effects of deep and moderate NMB on postoperative QOR in ambulatory gynecological laparoscopic surgery. We hypothesized that deep NMB improves postoperative QOR, compared to moderate NMB. The primary outcome was postoperative QOR in POD1. The secondary outcome was quality of surgical conditions, pain scores, time to meet PACU and hospital discharge, and opioid consumption

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II

Exclusion Criteria:

* Neuromuscular disorders

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | 24 hours postoperative
  Quality of recovery-40 (QoR-40) questionnaire, which includes five general quality of life dimensions: physical independence (5 items), pain (7 items), .emotional state (9 items), psychological support (7 items), and physical independence (5 items). Each item was graded with a 5-point score: none of the time, some of the time,usually, most of the time and all of the time. The total score on the QoR- 40 questionnaire ranges from 40 to 200 representing, respectively, extremely poor to excellent

SECONDARY OUTCOMES:
Postoperative pain | During the length of hospital stay post surgery (on average 24 hours)
  Visual analogue scale with its 0 to 10 score range: (0 (no pain) to 10 ( Severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Elite Medical Center, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
Web
Supporting Information: Study Protocol
Time Frame: 1 YEAR
Access Criteria: Web